CLINICAL TRIAL: NCT05760274
Title: Duration of Esophageal pH-impedance Measurement in Newborns and Infants With Suspected Gastroesophageal Reflux: 12 or 24 Hours?
Brief Title: Esophageal pH-MII Duration: 12 or 24 Hours?
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5080
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: multichannel intraluminal impedance and pH monitoring (MII/pH) — A pH-MII probe is inserted nasally into the esophagus, and the position verified by chest radiograph. pH-MII data are evaluated using manufacturer's software, and each tracing is manually reviewed and validated.

SUMMARY:
To check whether the first 12 hours of MII-pH recording are sufficient to diagnose gastroesophageal reflux disease (GERD) among newborns/infants, with a diagnostic accuracy similar to 24 hours of recording as currently advised.

DETAILED DESCRIPTION:
The results of the 24 hour MII-pH recording will be compared to those from the first 12 hour of the same study. To this end the study investigators will select the first 12 hour of the recording using the manufacturer's software (Diversatek Zvu Advanced GI Diagnostic Software). Published normal reference values will be used to confirm gastroesophageal reflux (GER). Appropriate statistical methods will be used to perform calculations. Subgroup analyses based on preterm birth, presence of bronchopulmonary dysplasia and type of prevalent GER symptom (respiratory or gastrointestinal) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 24 hours MII-pH performed for suspected GER

Exclusion Criteria:

* major malformations
* previous thoraco-abdominal surgery, gastrostomy, anti-GERD therapy (thickeners, alginates, H2 blockers, proton pump inhibitor - PPIs, etc.) in the 7 days preceding the MII-pH,
* ventilatory support (invasive or non-invasive) at the time of the MII-pH

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants 0-12 months who underwent 24 hour MII-pH for suspected GER
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
number of GER episodes | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
number of GER episodes reaching the proximal esophagus | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
time with pH<4 | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
bolus exposure index | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
bolus clearance time | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
symptom index | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
symptom association probability | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software

SECONDARY OUTCOMES:
number of GER episodes: subgroup analysis based on gestational age at birth, diagnosis of bronchopulmonary dysplasia (BPD), prevalent symptoms (respiratory or gastrointestinal) | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
number of GER episodes reaching the proximal esophagus: subgroup analysis based on gestational age at birth, diagnosis of BPD, prevalent symptoms (respiratory or gastrointestinal) | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
time with pH<4: subgroup analysis based on gestational age at birth, diagnosis of BPD, prevalent symptoms (respiratory or gastrointestinal) | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
bolus exposure index: subgroup analysis based on gestational age at birth, diagnosis of BPD, prevalent symptoms (respiratory or gastrointestinal) | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
bolus clearance time: subgroup analysis based on gestational age at birth, diagnosis of BPD, prevalent symptoms (respiratory or gastrointestinal) | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software
symptom index: subgroup analysis based on gestational age at birth, diagnosis of BPD, prevalent symptoms (respiratory or gastrointestinal) | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software. Range 0-100% (values ≥ 50% are significant).
symptom association probability: subgroup analysis based on gestational age at birth, diagnosis of BPD, prevalent symptoms (respiratory or gastrointestinal) | comparison between the first 12 hours of the test and the whole duration (24 hours)
  As detected by manufacturer's software. Range 0-100% (values ≥ 95% are significant).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nobile, MD, PhD, MSc, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nobile S, Rotunno G, Vandenplas Y, Salvatore S, Ummarino D, Quitadamo P, Aceti A, Vento G; GER12 Study Group. Assessing the Reliability of 12- vs 24-Hour Esophageal pH-Impedance Monitoring for Gastroesophageal Reflux in Infants. Am J Gastroenterol. 2025 Oct 13. doi: 10.14309/ajg.0000000000003796. Online ahead of print. PMID 41081569